CLINICAL TRIAL: NCT07383948
Title: Enhancing Parental Well-being in the NICU
Brief Title: Resilient Families Feasibility Trial
Acronym: R-FAM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Victoria A. Grunberg, PhD, Clinical Psychologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025P003422; 5K23HD110597-03 (NIH)
Record Dates: First submitted 2026-01-22; First posted 2026-02-03 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Parents
Keywords: Neonatal Intensive Care Unit; Parent Mental Health; Parent relationships

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- R-FAM Intervention (Other): A resiliency based intervention that includes 6-sessions with a clinician to help couples cope with the uncertainty and stress of the NICU admission.
  Interventions: Other: Resilient Families (R-FAM)
- Educational Program (Active Comparator): Participants will receive educational resources about adjusting to the NICU and coping with their stay.
  Interventions: Other: Educational Resources & Program

INTERVENTIONS:
Other: Resilient Families (R-FAM) — R-FAM is a resiliency intervention for couples with an infant admitted to the NICU. Parents will complete 6 guided sessions with a clinical psychologist that cover topics such as managing stress, staying in the present, and coping with uncertainty. Through these sessions, parents will learn skills to manage the "emotional roller-coaster" of the NICU, cope with stress, and connect with each other.
  Arms: R-FAM Intervention
Other: Educational Resources & Program — Parents will receive educational resources on how to cope with and adjust to the NICU stay.
  Arms: Educational Program

SUMMARY:
The goal of this study is to test the feasibility and acceptability of a dyadic, resiliency intervention ("Resilient Families;" R-FAM) that aims to reduce emotional distress and improve relationships among parents in the Neonatal Intensive Care Unit (NICU). To achieve this goal, the investigators are developing a randomized control trial where patients will be randomized to either the R-FAM condition or a minimally enhanced usual control (MEUC), which includes resources on parent mental health and coping in the NICU.

DETAILED DESCRIPTION:
The investigators aim to conduct a pilot feasibility randomized clinical trial (RCT) of R-FAM (Resilient Families) with NICU parents (up to N = 70 dyads) followed by a brief exit interview. The investigators will determine if the feasibility, acceptability, and fidelity of the program meet a priori benchmarks. The investigators also hope to establish preliminary efficacy that the program reduces parental emotional distress and other study outcomes described in sections below. The investigators will use qualitative data and data from the R-FAM open pilot to optimize the intervention and study procedures for future trials.

The investigators will conduct a single-blinded randomized clinical trial comparing the feasibility and acceptability of Resilient Families (R-FAM)-a resiliency intervention-with a one session educational program (minimally enhanced usual control) for parental couples ("dyads") of babies in the NICU. The investigators will also explore preliminary changes in outcomes and mechanisms to inform future trials. See Figure 1 for iterative development of R-FAM (the study is in years 3 and 4).

After enrollment, participants will be randomized to either the "Resilient Families" intervention or to the educational program (control). Dyads will be randomly assigned in a 1:1 ratio to intervention or control to ensure comparability between groups. The randomization schedule will be prepared using permuted blocks of size 2 and 4 by the unblinded study statistician and implemented in REDCap. All subjects will be given baseline psychological and behavioral assessments that will assess depression, anxiety, PTSD symptoms, and other psychological constructs.

ELIGIBILITY:
Inclusion Criteria:

* Adult parent/legal guardian (and/or their partner) of a baby admitted to the NICU within past week (age ≥ 18)
* Currently in an intimate relationship and will live with baby after NICU discharge
* At least one dyad member is emotionally distressed (GAD>=10 or PHQ >= 10)
* English fluency/literacy
* Ability and willingness to participate via live video

Exclusion Criteria:

* Baby is expected to pass away (as determined by medical team)
* Current, untreated psychosis or substance dependence/abuse
* Current self-report of suicidal ideation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Time Frame: Baseline to end of intervention (6 weeks)
  Level of anxiety endorsed on Hospital Anxiety & Depression Scale, from 0-21 with 21 indicating highest anxiety
Depression | Time Frame: Baseline to end of intervention (6 weeks)
  Level of depression endorsed on Hospital Anxiety & Depression Scale, from 0-21, with 21 indicating highest depression.
Posttraumatic Stress | Time Frame: Baseline to end of intervention (6 weeks)
  Level of posttraumatic stress endorsed on Impact of Event Scale-6, from 6-24 with 24 indicating highest posttraumatic stress

SECONDARY OUTCOMES:
Couple relationship functioning | Time Frame: Baseline to end of intervention (6 weeks)
  Couple satisfaction as reported on Couple Satisfaction Index, from 0-21 with 21 indicating highest couple satisfaction
Family Impact | Baseline to end of intervention (6 weeks)]
  Impact of child's illness as reported on Family Impact Scale, Revised, from 0-75 with 75 indicating lowest impact on family

CONTACTS AND LOCATIONS:
Overall Officials: Victoria A Grunberg, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Mass General Brigham, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No